CLINICAL TRIAL: NCT06835010
Title: Contradictory Effect of Sevoflurane and Dexmedetomidine on Kidney Function After Non-Cardiac Surgical Procedures Possibly Through Immunomodulation and Adjustment of Redox Milieu
Brief Title: Sevoflurane and Dexmedetomidine's Contrasting Renal Impacts After Non-Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Lotfy, Assistant Professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264PR666/4/24
Record Dates: First submitted 2025-02-09; First posted 2025-02-19 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: AKI - Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SEVO Group (Active Comparator)
  Interventions: Drug: Sevoflurane inhalant product
- DXM Group (Active Comparator)
  Interventions: Drug: Dexmedetomidine; Drug: Sevoflurane inhalant product

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine (Precedex, 100 µg/ml; Rewine Pharmaceutical; Varachha, Seurat, Gujarat) was administered before induction of anesthesia in the form of a 1 µg/kg; loading dose. The loading dose was diluted with 10 ml of normal saline and injected slowly for 10 minutes. IO infusion was prepared to provide 0.2-0.7 µg/kg/h, initially the lowest possible dose was infused and was increased gradually to control IO stress reflexes but with MAP, and HR monitoring to guard against IO hypotension and bradycardia. PO infusion was prepared to provide DXM in a dose of 0.15 µg/kg/h for 24-h. Placebo 0.9% saline solution was provided to patients of the SEVO group at a similar rate and duration.
  Arms: DXM Group
Drug: Sevoflurane inhalant product — Anesthesia was induced by fentanyl 1 μg/kg/min, propofol 1.5-2 mg/kg and rocuronium 0.5 mg/kg, then tracheal intubation was aided by gentle tracheal pressure and an endotracheal tube of appropriate size was inserted with the aid of fiberoptic laryngoscopy and patients were mechanically ventilated to keep ETCO2 in the range of 30-35 mmHg. Anesthesia was maintained for patients of both groups by sevoflurane 2% in oxygen 100% and rocuronium (0.15 mg/ kg) according to the requirements.

SUMMARY:
Postoperative acute kidney injury (PO-AKI) is a significant complication, especially after complex surgeries. The choice of anesthetic may influence PO-AKI risk. While sevoflurane (SEVO) has been associated with potential renal risks, dexmedetomidine (DXM) has demonstrated renoprotective effects in various surgical settings. These protective effects may be linked to DXM's immunomodulatory properties and influence on the redox balance. Given the common use of SEVO in major non-cardiac surgery and the potential for renal vulnerability, particularly in the elderly, this study hypothesizes that perioperative DXM infusion in patients undergoing major non-cardiac surgery with SEVO anesthesia will reduce the incidence and severity of PO-AKI, especially in those with pre-existing or borderline renal dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were assigned for TKR surgery;
* Patients with preoperative serum creatinine (SCr) levels of <1.1 mg/ml;
* Patients with controlled medical conditions;
* Patients free of exclusion criteria were enrolled in the study.

Exclusion Criteria:

* Male patients were excluded to guard against the impact of senile prostatic hypertrophy on kidney functions;
* Patients who had preoperative SCr of >1.1 mg/dl;
* Presence of any urological disorders, urological stone diseases;
* Patients with autoimmune diseases, medical disorders requiring maintenance on immunosuppressant therapy;
* Patients with cancer anywhere in the body were excluded.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Percentage Difference in Serum Creatinine levels After Dexmedetomidine Administration in Total Knee Replacement surgery under sevoflurane anesthesia. | 5 months
  The study assesses the mean percentage difference of serum creatinine levels in patients who was undergoing total knee replacement under sevoflurane anesthesia with Dexmedetomidine infusion (using standard laboratory assays).

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El Gharbyia, Egypt